CLINICAL TRIAL: NCT04175197
Title: The LegDeb2 Global Registry for the Treatment of Superficial Femoral, Popliteal or Below-The-Knee Artery Lesions Using the Legflow DrugEluting Balloon
Brief Title: LegDeb2 Global Registry for Use of Legflow in Peripheral Arteries
Acronym: LEGDEB2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Eugenio Stabile, Associate Professor of Cardiovascular Medicine, Federico II University
Other Study IDs: LEGDEB2 v.3.1
Record Dates: First submitted 2019-11-12; First posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Peripheral Arterial Disease; Superficial Femoral Artery Stenosis; Iliac Artery Stenosis; Arterial Occlusive Diseases; Popliteal Artery Stenosis; Critical Limb Ischemia
Keywords: Stenosis; Drug Coated Balloon; Paclitaxel; Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease; Arterial Occlusive Diseases; Chronic Limb-Threatening Ischemia; Constriction, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Cohort: Subjects with symptoms of intermittent claudication and/or critical limb ischemia (Rutherford Class 2-3-4-5-6) with angiographic evidence of femoropopliteal-below-the-knee arterial occlusion or stenosis
  Interventions: Device: Drug Coated Balloon

INTERVENTIONS:
Device: Drug Coated Balloon — Legflow Drug Coated Balloon

SUMMARY:
LEGDEB2 is a Global Registry for the Treatment of Superficial Femoral and/or Popliteal or Below-The-Knee or Iliac Artery Lesions Using the Legflow Drug-Eluting Balloon

DETAILED DESCRIPTION:
LEGDEB2 is a Global Registry aimed to prospectively collect and assess global safety and efficacy data on the Legflow Drug Eluting Balloon (DEB) in treatment of atherosclerotic disease of the superficial femoral and/or popliteal and/or below-the-knee and/or iliac arteries in "real world" patient population.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years or minimum age as required by local regulations.

* Subject with documented diagnosis of lower extremities arterial disease (LEAD).
* Angiographically documented single or multiple lesions/occlusions (de novo or re-stenotic lesion(s) or in-stent restenosis within the target vessels with a minimum lesion length of 2 cm including bilateral disease if both limbs are treated within 35 days.
* Positive diagnostic indication for PTA with a DEB in accordance with the Instructions For Use (IFU) of the Legflow DEB.
* Adequate distal run-off to the ankle (at least one native calf vessel [posterior tibial, anterior tibial, or peroneal arteries] is patent, defined as ≤ 50% diameter stenosis) either pre-existing or successfully re- established prior to target lesion treatment.
* Adequate inflow (≤ 50% diameter stenosis) either pre-existing or successfully re-established prior to target lesion treatment.
* Female subjects of childbearing potential must have a negative pregnancy test ≤ 7 days before enrollment.
* Signed and dated Patient Informed Consent (PIC) form.
* Ability and willingness to comply with the clinical investigation plan (CIP).
* Life expectancy, in the Investigator's opinion, of at least 12 months

Exclusion Criteria:

* High probability of non-adherence to CIP follow-up requirements.
* Failure to successfully cross the target lesion with a guide wire (successful crossing means tip of the guide wire distal to the target lesion in the absence of flow limiting dissections or perforations).
* Lesion within or adjacent to an aneurysm or presence of a popliteal aneurysm.
* Acute or sub-acute thrombus in the target vessel.
* Target lesion also requires treatment with alternative drug eluting technology-based therapy or other antiproliferative therapy (cryoplasty, brachytherapy).
* Plan for surgical or interventional procedure within 30 days after the study procedure (except for bilateral target limb treatment).
* Known allergies or sensitivities to heparin, aspirin, other anti- coagulant/anti-platelet therapies, and/or paclitaxel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with symptoms of intermittent claudication and/or critical limb ischemia (Rutherford Class 2-3-4-5-6) with angiographic evidence of femoropopliteal-below-the-knee iliac arterial occlusion or stenosis will be consecutively screened and enrolled based on the study inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 512 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Freedom from Clinically driven TLR | 12 Months
  Freedom from clinically-driven target lesion revascularization (TLR) within 12 months post-index procedure, which is defined as:
  * Any re-intervention within the target lesion(s) due to symptoms
Safety: Freedom from MAE | 30 days
  A composite of freedom from device- and procedure-related mortality through 30 days, freedom from device or procedure related mortality, freedom from any cardiac or cardiovascular death, freedom from major target limb amputation

SECONDARY OUTCOMES:
Freedom from MALE and MACCE | 30 days, 6 Months, 12 Months, 24 Months, 36 Months
  MALE is defined as acute limb ischemia, urgent revascularization or mayor amputation of the treated limb MACCE is defined as Death, Acute myocardial infarction or stroke
Freedom from all cause mortality | 30 days, 6 Months, 12 Months, 24 Months, 36 Months
  all cause mortaliy
Freedom from CD-TLR | 24 Months, 36 Months
  Clinically driven Target Lesion Revascularization
Freedom from CD-TVR | 6 Months, 12 Months, 24 Months, 36 Months
  Clinically driven Target Vessel Revascularization Clinically-driven TVR is defined as any re-intervention within the target vessel due to symptoms
Freedom from Major target limb amputation | 30 days, 6 Months, 12 Months, 24 Months, 36 Months
  Major target limb amputation
Primary sustained clinical improvement | 6 Months, 12 Months, 24 Months, 36 Months
  Primary sustained clinical improvement is defined as sustained upward shift of at least 1 category on Rutherford classification as compared to baseline without the need for repeated TLR or surgical revascularization in amputation-free surviving subjects
Device Success | Day 1
  Device success is defined as successful delivery, balloon inflation and deflation and retrieval of the intact study device without burst below the rated burst pressure (RBP).
Procedural Success | Day 1
  Procedural success is defined as residual stenosis of ≤ 50% (non-stented subjects) or ≤ 30% (stented subjects) by visual estimate
Clinical Success | Day 1
  Clinical success is defined as procedural success without in hospital MALE and/or MACCE

CONTACTS AND LOCATIONS:
Locations (7):
- Italy (3):
  - Policlinico di Monza, Monza
  - Università Federico II - Dipartimento Scienze Biomediche Avanzate, Napoli
  - Policlinico Umberto I, Roma
- Mexico (4):
  - Angeles del Carmen, Guadalajara
  - Consulta Privada Cardiovascular Research Institute, Guadalajara
  - Hospital Angeles Mocel, Mexico City
  - Hospital Lopez Mateos, Mexico City

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Stabile E, Gerardi D, Magliulo F, Zhelev D, Chervenkoff V, Taeymans K, Kotasov D, Goverde P, Giugliano G, Trimarco B, Esposito G. One-Year Clinical Outcomes of the Legflow Drug-Coated Balloon for the Treatment of Femoropopliteal Occlusions Registry. J Endovasc Ther. 2019 Feb;26(1):26-30. doi: 10.1177/1526602818823557. PMID 30760132